CLINICAL TRIAL: NCT03402659
Title: A Double-Blind, Placebo-Controlled Proof-of-Concept Study of a Selective p38 MAP Kinase Alpha Inhibitor, Neflamapimod, Administered for 24 Weeks in Subjects With Mild Alzheimer's Disease
Brief Title: Proof-of-Concept Study of a Selective p38 MAPK Alpha Inhibitor, Neflamapimod, in Subjects With Mild Alzheimer's Disease
Acronym: REVERSE-SD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: Worldwide Clinical Trials (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP-VX17-745-304
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — VX-745

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neflamapimod (Experimental): 40 mg hard gelatin capsules, taken twice daily with food.
  Interventions: Drug: neflamapimod
- placebo (Placebo Comparator): hard gelatin capsules containing excipients only, weight- and size-matched; taken twice daily with food.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: neflamapimod — 40 mg neflamapimod capsule
  Other Names: VX-745
  Arms: neflamapimod
Other: placebo — matching placebo capsule
  Arms: placebo

SUMMARY:
This is a phase 2b, double-blind, placebo controlled proof-of-concept study of a an oral small molecule selective inhibitor of p38 alpha kinase, neflamapimod, administered for 24 weeks in subjects with mild Alzheimer's disease. The primary objective is to demonstrate significant improvement relative to placebo-treatment in episodic memory function, as assessed by the Hopkins Verbal Learning Test. Secondary endpoints include Clinical Dementia Rating scale (CDR), Wechsler Memory Scale (WMS), Mini-Mental-Status-Examination (MMSE) and Cerebrospinal fluid (CSF) biomarkers of AD disease activity and progression.

DETAILED DESCRIPTION:
Details provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 55 to 85 years, inclusive.
2. Willing and able to provide informed consent.
3. Must have mild cognitive impairment (MCI) or mild AD with evidence of progression ("Mild-AD"), as defined by the following:

   1. CDR-Global Score of 0.5 or 1.0, with CDR memory subscore of at least 0.5.
   2. MMSE score ranging from 20 to 28, inclusive.
   3. Positive biomarker for AD, as defined by a CSF Aβ1-42R below the threshold and phospho-tau above the threshold for the assay utilized in the study and assessed by the central laboratory.
4. Computed tomography (CT) or magnetic resonance imaging (MRI) findings within 2 years of Screening that are compatible with AD and no other pathologic processes that might potentially account for the subject's cognitive impairment.
5. If the subject is taking a single drug for AD (e.g., donepezil or other cholinesterase inhibitors or memantine; dual therapy is excluded), he/she has been on a stable dose for at least 2 months prior to baseline, and the dose must remain unchanged during the study unless required for management of adverse events (AEs).
6. Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.
7. Must have reliable informant or caregiver.

Exclusion Criteria:

1. Evidence that the primary basis for cognitive impairment is neurodegenerative disease other than AD, including, but not limited to, vascular dementia, dementia with Lewy bodies, and Parkinson's disease.
2. Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
3. History of major and active psychiatric disorder, moderate to severe depressive symptoms, and or other concurrent medical condition that, EIP-VX17-745-304, Version 1.0, 17 November, 2017 Page 7 of 46 EIP Pharma, LLC Confidential in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
4. Diagnosis of alcohol or drug abuse within the previous 2 years.
5. History of cancer within the last 5 years, except basal cell carcinoma, squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
6. Poorly controlled clinically significant medical illness.
7. History of serum B12 abnormality, anemia with hemoglobin ≤10 g/dL, thyroid function abnormality, electrolyte abnormality, or positive syphilis serology that have not been corrected and/or otherwise addressed.
8. History of epilepsy or unexplained seizure within the past 5 years.
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 × the upper limit of normal (ULN), total bilirubin >2 × ULN, and/or International Normalized Ratio (INR) >1.5
10. Known human immunodeficiency virus, hepatitis B, or active hepatitis C virus infection.
11. Subject participated in a study of an investigational drug less than 3 months or 5 half-lives of the investigation drug, whichever is longer, before enrollment in this study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Alam, MD, Study Director — EIP Pharma
Locations (38):
- United States (16):
  - Alliance for Research, Long Beach, California
  - Pacific Research Network, San Diego, California
  - CITrials, Santa Ana, California
  - Southern California Research, LLC, Simi Valley, California
  - Viking Clinical Research, Temecula, California
  - Miami Dade Medical Research Institute, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - MassGeneral Institute for Neurodegenerative Disease, Charlestown, Massachusetts
  - Manhattan Behavioral Medicine, New York, New York
  - Alzheimer's Memory Center and Research Institute, Charlotte, North Carolina
  - Northwest Clinical Research Center, Seattle, Washington
- Czechia (5):
  - Neuro HK, s.r.o. POLIKLINIKA CHOCEŇ, a.s., Choceň
  - Cerebrovaskulární poradna s.r.o., Moravská Ostrava
  - Clintrial S.R.O, Prague
  - Private Psychiatric Centre, Prague
  - Vestra Clinics S.R.O, Rychnov nad Kněžnou
- Denmark (3):
  - CCBR Clinical Research, Aalborg, Aalborg
  - CCBR Clinical Research, Ballerup, Ballerup Municipality
  - CCBR Clinical Research, Vejle, Vejle
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Alzheimer Research Center, Amsterdam
  - Amphia Ziekhuis, Breda
- United Kingdom (11):
  - MAC Clinical Research Tankersley, Barnsley
  - Re:Cognition Health Birmingham, Birmingham
  - MAC Clinical Research Blackpool, Blackpool
  - Fulbourn Hospital, Cambridge
  - MAC Clinical Research Leeds, Leeds
  - MAC Clinical Research Liverpool, Liverpool
  - Re:Cognition Health London, London
  - St. Pancras Clinical Research, London
  - MAC Clinical Research Manchester, Manchester
  - Re:Cognition Health Plymouth, Plymouth
  - 5 Boroughs/North West Boroughs Healthcare NHS Foundation Trust, Warrington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prins ND, Harrison JE, Chu HM, Blackburn K, Alam JJ, Scheltens P; REVERSE-SD Study Investigators. A phase 2 double-blind placebo-controlled 24-week treatment clinical study of the p38 alpha kinase inhibitor neflamapimod in mild Alzheimer's disease. Alzheimers Res Ther. 2021 May 27;13(1):106. doi: 10.1186/s13195-021-00843-2. PMID 34044875
- [Derived] Tormahlen NM, Martorelli M, Kuhn A, Maier F, Guezguez J, Burnet M, Albrecht W, Laufer SA, Koch P. Design and Synthesis of Highly Selective Brain Penetrant p38alpha Mitogen-Activated Protein Kinase Inhibitors. J Med Chem. 2022 Jan 27;65(2):1225-1242. doi: 10.1021/acs.jmedchem.0c01773. Epub 2021 May 11. PMID 33974419

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Arm of trial including the 83 subjects that were randomly assigned (1:1) to take placebo
- Neflamapimod Arm: Arm of trial including the 78 subjects that were randomly assigned (1:1) to take neflamapimod (active study drug).
Period: Overall Study
Arm/Group | Placebo Arm | Neflamapimod Arm
Started | 83 | 78
Completed | 78 | 73
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Neflamapimod Arm | Total
Number analyzed (Participants) | 83 | 78 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 69 | 62 | 131
Age, Continuous [Mean (Full Range); unit: years] | 72.6 [56 to 85] | 70.8 [56 to 84] | 71.8 [56 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 80
  Male | 40 | 41 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 79 | 77 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 10 | 10 | 20
  United States | 38 | 35 | 73
  Czechia | 3 | 6 | 9
  Denmark | 3 | 4 | 7
  United Kingdom | 29 | 23 | 52
Weight [Mean (Full Range); unit: Kg] | 74.4 [45 to 111] | 75.6 [48.9 to 161] | 75 [45 to 161]

OUTCOME MEASURES:

1. Primary Outcome: Total and Delayed Recall on the Hopkins Verbal Learning Test - Revised (HVLT-R)
Description: Combined change from baseline in z-scores of total and delayed recall on the Hopkins Verbal Learning Test - Revised (HVLT-R) in neflamapimod-treated subjects compared to placebo. The primary endpoint was analyzed using Mixed Model for Repeated Measures (MMRM) with fixed effects for treatment, background AD-specific therapy, CDR-Global Score of 0.5 versus 1.0, scheduled visit (nominal) and scheduled visit by treatment interaction, random effect for subject and baseline Z-score as a covariate.
  For baseline total and delayed recall, a z-score for each subject is defined by z=(x-m)/s where x is the subject's recall at baseline, and m and s are the overall mean and overall standard deviation of recall at baseline across all subjects. A composite baseline z-score for each subject is calculated using equal weighting in the following way: Z=0.5*z-score for total recall at baseline + 0.5*z-score for delayed recall at baseline. For HVLT-R, higher score indicates improvement.
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 72 | 71
Z-score | -0.09679 (0.074840) | -0.15776 (0.085805)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.564, Mixed Models Analysis; Mean Difference (Final Values) = -0.06098, 95% CI 2-sided [-0.26973 to 0.14777], Standard Error of Mean 0.105548

2. Secondary Outcome: Wechsler Memory Scale (WMS) Immediate and Delayed Recall
Description: Change from baseline in Wechsler Memory Scale(WMS) immediate and delayed recall composites in neflamapimod-treated subjects compared to placebo. WMS scores were analyzed using Mixed Model for Repeated Measures (MMRM) with fixed effects for treatment, background AD-specific therapy, CDR-Global Score of 0.5 versus 1.0, scheduled visit (nominal) and scheduled visit by treatment interaction, random effect for subject and baseline Z-score as a covariate. Composite scores for immediate and delayed recall are the combination of all immediate and delayed recall task raw scores and ranges from 0-228. A higher score indicates improvement.
  The following tests in WMS are done both for immediate and delayed recall: Logical Memory test, in which subject is read a story; Verbal-Paired Associates, in which subject is given pairs of words and asked remember which words go together; and Visual Reproduction, in which subject is given drawings of specific shapes
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 77 | 71
Scores on a scale | 16.6 (2.09) | 16.0 (2.07)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.823, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-6.0 to 4.8], Standard Error of Mean 2.72

3. Secondary Outcome: Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB)
Description: Change from baseline in total score of Clinical Dementia Rating Scale - Sum of Boxes (range 0-18) in neflamapimod-treated subjects compared to placebo. CDR-SB scores were analyzed using Mixed Model for Repeated Measures (MMRM) with fixed effects for treatment, background AD-specific therapy, CDR-Global Score of 0.5 versus 1.0, scheduled visit (nominal) and scheduled visit by treatment interaction, random effect for subject and baseline Z-score as a covariate. CDR-SB score is calculated by adding the individual scores from 6 domains, Memory, Orientation, Judgement and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care. CDR-SB scores range from 0-18, where a lower score indicates improvement. The scale is administered in a semi-structured interview format with both the patient and the caregiver/informant.
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 78 | 74
Scores on a scale | 1.0 (0.20) | 1.1 (0.21)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.806, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.6], Standard Error of Mean 0.25

4. Secondary Outcome: Mini-Mental State Examination (MMSE)
Description: Changes from baseline in Mini-Mental State Examination (MMSE) scores were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value. The MMSE is scored from 0-30 with a higher score indicating improvement. The MMSE includes questions that test orientation, attention, memory, language and visual-spatial skills.
Time Frame: Baseline and 26 Weeks (Follow-up visit, 2 weeks from end of dosing)
Population: All participants who had analyzable results at Baseline and Follow-up Visit (2 weeks post-treatment)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 79 | 70
Scores on a scale | -0.5 (0.31) | -0.8 (0.33)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.489, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.39

5. Secondary Outcome: Cerebrospinal Fluid Total Tau
Description: Change from, baseline in Total Tau (t-tau) were compared using an ANCOVA with treatment group, background ADspecific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants with analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 10.0 (6.83) | -8.6 (7.36)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.031, ANCOVA; Mean Difference (Final Values) = -18.8, 95% CI 2-sided [-35.8 to -1.8], Standard Error of Mean 8.60

6. Secondary Outcome: Cerebrospinal Fluid Phospho-tau
Description: Change from baseline in Phospho-Tau (p-tau181) were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 0.9 (0.63) | -1.1 (0.68)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.012, ANCOVA; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.6 to -0.5], Standard Error of Mean 0.79

7. Secondary Outcome: Cerebrospinal Fluid Amyloid Beta 1-40
Description: Change from baseline in Amyloid beta (AB1-40) were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 399.7 (249.18) | 282.3 (268.58)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.709, ANCOVA; Mean Difference (Final Values) = -117.4, 95% CI 2-sided [-738.9 to 504.2], Standard Error of Mean 314

8. Secondary Outcome: Cerebrospinal Fluid Amyloid Beta 1-42
Description: Change from baseline in Amyloid beta (AB1-42) were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants who had analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 31.1 (12.70) | 10.0 (13.75)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.192, ANCOVA; Mean Difference (Final Values) = -21.0, 95% CI 2-sided [-52.7 to 10.7], Standard Error of Mean 16.03

9. Secondary Outcome: Cerebrospinal Fluid Neurogranin
Description: Change from baseline in Neurogranin were compared using an ANCOVA with treatment group, background ADspecific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants with analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 11.1 (9.16) | -9.9 (9.82)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.068, ANCOVA; Mean Difference (Final Values) = -21.0, 95% CI 2-sided [-43.6 to 1.6], Standard Error of Mean 11.43

10. Secondary Outcome: Cerebrospinal Fluid Neurofilament Light Chain
Description: Change from baseline in Neurofilament Light Chain (NFL) were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants with analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
pg/mL | 231.9 (61.31) | 121.7 (66.92)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.156, ANCOVA; Mean Difference (Final Values) = -110.1, 95% CI 2-sided [-262.7 to 42.4], Standard Error of Mean 77.11

11. Secondary Outcome: Cerebrospinal Fluid P-tau/AB1-42 Ratio
Description: Changes in the ratio of Phospho-Tau/Amyloid Beta (p-tau181/AB1-42) were compared using an ANCOVA with treatment group, background AD-specific therapy, CDR-Global Score as main effects and the baseline assessment as the covariate. The results of the ANCOVA are summarized using the treatment groups' least square means, the difference between the treatment groups' least square means, the 95% confidence interval for the treatment group difference and the p-value.
Time Frame: Baseline and 24 weeks
Population: All participants with analyzable results at Baseline and Week 24
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo Arm | Neflamapimod Arm
Number analyzed (Participants) | 68 | 62
ratio | -0.0 (0) | -0.0 (0)
Statistical Analysis 1: Comparison: Placebo Arm vs Neflamapimod Arm; Mean change from baseline neflamapimod vs placebo; Test type: Other; p = 0.590, ANCOVA; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.0 to 0.0], Standard Error of Mean 0

ADVERSE EVENTS:
Time Frame: Up to 29 weeks. AEs occurring from when the subject signed the ICF until up to 30 days after the last dose were collected. Any AEs occurring before the start of treatment (i.e., before the first dose of the investigational product) were recorded in the medical history.
Description: Any sign, symptom, or disease present before starting the treatment period were only considered AEs if they worsen after starting the treatment period.
Arm/Group | Placebo Arm | Neflamapimod Arm
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/78
Serious Adverse Events (participants affected / at risk) | 3/83 | 2/78
Other Adverse Events (participants affected / at risk) | 16/83 | 18/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=83) | Neflamapimod Arm (N=78)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Multiple Myeloma occurred in one subject. It was not considered related to neflamapimod.
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — One SAE of Hypokalemia was reported. It was considered not related to neflamapimod.
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=83) | Neflamapimod Arm (N=78)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (8) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 4 (6) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03402659/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03402659/SAP_001.pdf